CLINICAL TRIAL: NCT02578303
Title: Association Between Cerebral Arterial Vascular Flow and Sleep Apnea in Neurodegenerative Alterations
Acronym: VAAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital Saint Quentin (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RCB / N° 2014-A01617-40
Record Dates: First submitted 2015-10-09; First posted 2015-10-16 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2019-07

CONDITIONS: Alzheimer Disease
Keywords: sleep apnea; phase-contrast MRI; cerebral blood flow; vascular risk factor; dementia
MeSH Terms: conditions — Alzheimer Disease; Sleep Apnea Syndromes; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dementia group (Experimental): Assessed by the insertion of an interaction parameter between cerebral blood flow and the group label(dementia or no-dementia).
  ROC method will be used to find a threshold value of IAH that separates the two groups.
  Interventions:
  * Vascular flow measurement by PC-MRI
  * Neuropsychological assessment
  * Registration of sleep apnea
  * Registration of blood pressure
  * ECG holters
  * Blood test
  * Geriatric standard evaluation
  Interventions: Other: Vascular flow measurement by PC-MRI
- control group (Other): Assessed by the insertion of an interaction parameter between cerebral blood flow and the group label(dementia or no-dementia).
  ROC method will be used to find a threshold value of IAH that separates the two groups.
  Interventions:
  * Vascular flow measurement by PC-MRI
  * Neuropsychological assessment
  * Registration of sleep apnea
  * Registration of blood pressure
  * ECG holters
  * Blood test
  * Geriatric standard evaluation
  Interventions: Other: Vascular flow measurement by PC-MRI

INTERVENTIONS:
Other: Vascular flow measurement by PC-MRI — participants will undergo vascular flow measurement by PC-MRI at intra and extracranial levels

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is a sleep-disordered breathing characterized by the occurrence of repeated upper airway obstructions leading to airflow reduction (hypopnea) or cessation (apnea). The apnea-hypopnea index (AHI) is the number of apneas and hypopneas per hour of sleep. OSA patients often report cognitive complaints.

About 25% of the elderly population is affected by this syndrome with a drastic increase of this rate among dementia patients. OSAS is considered to be an important risk factor for the development of hypertension, heart disease and stroke.

DETAILED DESCRIPTION:
Numerous studies pointed out the close relationship between sleep apnea and cognitive impairment. To the investigators' knowledge, no trials have assessed the existence of a relationship between the IAH index and the cerebral arterial blood flow rate (macrocirculation). Developments in magnetic resonance imaging (MRI) provide new insights into the quantitative study of blood flow through phase contrast MRI also called "flow MRI". The main hypothesis tested in this study is the existence of a relationship between OSAS and total cerebral arterial vascular inflow measured by PC-MRI (in mL/min) in the elderly population.

* Primary outcome: The apnea/hypopnea index (measured by nocturnal respiratory polygraphy) and total arterial flow rate (measured by PC-MRI)
* Secondary outcomes:

  1. Measurement of arrhythmia
  2. Measurement of arterial blood pressure

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients about or over 75 years
2. Any gender
3. Dementia Group:

   3.1. MMSE (Mini Mental State Examination)> 15

   3.2. Diagnosis of dementia established according to DSM-IV

   3.3. Dementia of the Alzheimer type from NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association)
4. Control Group:

   Preserved cognitive function corresponding to a normal MMSE score by the standards of Poitrenaud
5. Ability to understand and give consent freely (for demented subjects, a legal representative will be delegate)

Exclusion Criteria:

1. Elderly patients under 75 years
2. Anyone with a classic contraindication to MRI

   2.1 Major behavioral disorders that do not allow the realization of MRI in optimal conditions

   2.2 Claustrophobia

   2.3 Presence of foreign non-compliant material

   2.4 Presence of intraocular metal body
3. Having a history of chest surgery or neurosurgical
4. Chronic respiratory failure
5. Suffering from dementia other than that associated with Alzheimer's disease
6. Patients with a handicap
7. Patients under legal protection

Ages: 75 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2015-05; Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Total arterial flowrate (measured by PC-MRI debit ml/Mn) | at day 1 after inclusion

SECONDARY OUTCOMES:
sleep apnea measured by elderly polygraphy (Number of apneas / night) | at day 1 after inclusion up to 24 heures

CONTACTS AND LOCATIONS:
Overall Officials: ATTIER Jadwiga, MD, Principal Investigator — CH SAINT-QUENTIN
Locations (1):
- CH Saint-Quentin, Saint-Quentin, France

IPD SHARING:
Plan to Share IPD: No